CLINICAL TRIAL: NCT03778684
Title: Impact of Obesity on Intracytoplasmic Sperm Injection Cycle Outcome: a Prospective Cohort Study
Brief Title: Obesity and Intracytoplasmic Sperm Injection Cycle Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Ahmad Mohamed Makhlouf, Assistant Lecturer, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ICSI-Alaa
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Body Mass Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Body mass index without central obesity (Experimental)
  Interventions: Diagnostic Test: Visceral fat thickness; Diagnostic Test: Body mass index
- High Body mass index with central obesity (Experimental)
  Interventions: Diagnostic Test: Visceral fat thickness; Diagnostic Test: Body mass index

INTERVENTIONS:
Diagnostic Test: Visceral fat thickness — An initial longitudinal sweep will be done from the xiphoid process to the umbilicus to determine the area of maximum pre-peritoneal fat thickness.
Diagnostic Test: Body mass index — Weight and height will be measured with subjects in a standing position wearing light clothes and no shoes.

SUMMARY:
Obesity has been associated with menstrual irregularities, chronic an-ovulation, infertility, and poor outcomes in women undergoing in vitro fertilization.

There is strong evidence that obesity is associated with a higher n vitro fertilization cycle cancellation rate (despite administration of higher doses of exogenous gonadotrophins), a lower mature oocyte yield and lower number of cryopreservation cycles.

Furthermore, obese women have been shown to have impaired response to ovarian stimulation and significantly lower live births after in vitro fertilization. Indeed, obesity affects many ovarian intra-follicular steroidogenic, metabolic and inflammatory pathways.This is particularly evident in women with abdominal (central obesity). Waist circumference measurement is used to identify individuals with abdominal obesity but it cannot differentiate between intra-abdominal fat and subcutaneous abdominal fat accumulation.

The reliable measurement of visceral fat and subcutaneous fat is not only important as a tool to predict cardiovascular and metabolic disease risk, but it is also essential to evaluate the effect of these fat compartments on female reproductive function. Intra-abdominal fat accumulation is related to insulin resistance in women with polycystic ovary syndrome and in these women the resulting hyperinsulinemia contributes to an-ovulation.

Obese anovulatory women with polycystic ovary syndrome who resume ovulation during a 6-month lifestyle program lose more visceral fat with no difference in the change of subcutaneous fat compared to the women who did not resume ovulation.

Another recent study that enrolled 140 non-polycystic ovary syndrome in vitro fertilization women demonstrated that women with increased waist circumference and higher follicular fluid leptin have less oocytes fertilized and failed in vitro fertilization outcomes. Increased intra-abdominal fat during early pregnancy is associated with insulin resistance and increased diastolic blood pressure and it can predict glucose intolerance in later pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age of women 18 - 35 yrs old.
* Women with Body mass index I 18 - 35 kg/m2.
* Infertile women with an indication for In vitro fertilization
* Anticipated normal responders.
* Normal uterine cavity by trans-vaginal ultrasound.

Exclusion Criteria:

* Poly cystic ovarian syndrome
* Diabetic patients.
* Known Poor ovarian response
* Patients with abnormal uterine cavity.
* Refusal to participate in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-11-26 (Actual)

PRIMARY OUTCOMES:
Number of women will be pregnant (clinical pregnancy rate) | 1 month
  a pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided